CLINICAL TRIAL: NCT06210529
Title: A Single-center, Prospective Clinical Study of High-intensity Focused Ultrasound Tumor Treatment System(Super Knife) in the Treatment of Breast Cancer
Brief Title: Clinical Study of High-intensity Focused Ultrasound Tumor Treatment System(Super Knife) in the Treatment of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN 10
Record Dates: First submitted 2024-01-02; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (treatmen once) (Experimental)
  Interventions: Device: a high-intensity focused ultrasound tumor treatment system (Super Knife)
- Group B (treatmen twice) (Experimental)
  Interventions: Device: a high-intensity focused ultrasound tumor treatment system (Super Knife)

INTERVENTIONS:
Device: a high-intensity focused ultrasound tumor treatment system (Super Knife) — All participants will be randomly divided into groups A and B. Participants in group A will receive a high-intensity focused ultrasound tumor treatment (Super Knife) once, and participants in group B will receive treatment twice (4 weeks, one cycle).. Breast cancer surgery was performed at 3 months ± 1 week after the Super Knife treatment.

SUMMARY:
Breast cancer is the most common cancer diagnosed among women and is the second leading cause of cancer death among women after lung cancer. The treatment methods of breast cancer include surgery, chemotherapy, radiotherapy and so on. The investigators discover a High-intensity focused ultrasound therapy to treat breast tumor, which is a non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

ECOG Performance Status of 0-1; Histological confirmed invasive breast cancer; Breast cancer tumor measuring ≥2 cm in maximal diameter and a single lesion as measured by mammogram, breast ultrasound, or breast MRI; Breast tumor's borders from the skin are greater than 1 cm; No lymph node or distant metastasis; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, Platelets ≥ 50 × 109/L, Hemoglobin ≥ 9.0 g/dl iv; Serum creatinine ≤1.5 x upper limit of normal (ULN); AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN; Left ventricular ejection fraction ≥ 50%.

Exclusion Criteria:

Inflammatory breast cancer, bilateral breast cancer, or occult breast cancer; Any kind of prior treatment for breast cancer, including chemotherapy, radiotherapy, endocrine therapy and so on; Pregnant and lactating women; Patients who have participated in other clinical trials.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 1 month after surgery
  pCR is defined as the absence of residual invasive cancer in the breast and the lymph nodes.

SECONDARY OUTCOMES:
Disease control rate | In the first month, the second month, the third month
  The percentage of patients whose therapeutic intervention has led to a complete response, partial response, or stable disease.
Objective response rate | In the first month, the second month, the third month
  The percentage of patients whose therapeutic intervention has led to a complete response, partial response.
Adverse events | 1 month after surgery
  Adverse events during and after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No